CLINICAL TRIAL: NCT03357172
Title: Determination of Factors Involved in the Regulation of Immune Responses After Allogeneic Hematopoietic Stem Cell Transplantation
Acronym: REAL-GREFFE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2018-A03267-48
Record Dates: First submitted 2017-11-24; First posted 2017-11-29 (Actual); Last update posted 2019-10-14 (Actual); Status verified 2019-10

CONDITIONS: Allogeneic Hematopoietic Stem Cell Transplantation
Keywords: Immune recovery; Immunomodulatory cells; GVHD; GVL
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Recipient (Experimental)
  Interventions: Biological: Blood Sample; Biological: Bone marrow aspiration
- Donor (Experimental)
  Interventions: Biological: Blood sample; Biological: Allogeneic hematopoietic stem cell sample

INTERVENTIONS:
Biological: Blood Sample — Additional blood sample before graft, D0, D7, D15, D21, D30, D60, D90, D180, Y1, Y2
  Arms: Recipient
Biological: Bone marrow aspiration — Additional bone marrow aspiration before graft, D30, D90, Y1
  Arms: Recipient
Biological: Blood sample — Before donation
  Arms: Donor
Biological: Allogeneic hematopoietic stem cell sample — Allogeneic hematopoietic stem cell sample
  Arms: Donor

SUMMARY:
The study concerns donors and patients receiving allogeneic stem cell haematopoietic transplantation. The aim of the study is to analyse HSC graft content in immune effector T (naive, memory, activated, exhausted) and immunoregulatory cell subtypes (Tregs, iNKT, MDSC) and correlate the results with post-transplant immune reconstitution of those different cell subtypes and clinical events (graft-versus-host-disease, relapse, infections). An ancillary study will focus on the impact of microbiota dysbiosis on post-transplant immune response and regulatory cell subsets.

ELIGIBILITY:
Inclusion Criteria:

* patient of the Nancy CHRU, for whom a CSH allograft is planned. or
* hematopoietic stem cell donors received at Nancy's CHRU for the duration of the research

Exclusion Criteria:

* Positive HIV
* active hepatitis B or C infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 700 (Estimated)
Dates: Start 2019-10-01 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Proportions of regulatory immune cells in peripheral blood. | After 7 days, 15 days, 21 days, 30 days, 60 days, 90 days, 180 days, 1 year, 2 years

SECONDARY OUTCOMES:
Occurrence of graft versus host (GVH) reaction after allografting of CSH | After 7 days, 15 days, 21 days, 30 days, 60 days, 90 days, 180 days, 1 year, 2 years
Incidence of relapse | After 7 days, 15 days, 21 days, 30 days, 60 days, 90 days, 180 days, 1 year, 2 years
Incidence of infections | After 7 days, 15 days, 21 days, 30 days, 60 days, 90 days, 180 days, 1 year, 2 years
Progress-free survival | After 7 days, 15 days, 21 days, 30 days, 60 days, 90 days, 180 days, 1 year, 2 years
Overall survival | After 7 days, 15 days, 21 days, 30 days, 60 days, 90 days, 180 days, 1 year, 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- CHRU de Nancy, Vandœuvre-lès-Nancy, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Notarantonio AB, Morisset S, Piucco R, Peres M, Boulange L, Alitcher A, Brouard J, Monchablon L, Campidelli A, El Ouahabi S, Guisnel C, Moulin C, Kicki C, Roth-Guepin G, Feugier P, Bittencourt MC, Aarnink A, D'Aveni-Piney M, Hergalant S, Pagliuca S, Rubio MT. Differential Clinical and Immunological Impacts of Anti-T-Lymphocyte Globulin (ATLG) vs. Anti-Thymocyte Globulin (ATG) in Preventing Graft-Versus-Host Disease Post-Allogeneic Hematopoietic Stem Cell Transplantation: A Comparative Study. Am J Hematol. 2025 Apr;100(4):626-637. doi: 10.1002/ajh.27619. Epub 2025 Feb 4. PMID 39905816
- [Derived] Notarantonio AB, Bertrand A, Piucco R, Fievet G, Sartelet H, Boulange L, de Isla N, De Carvalho Bittencourt M, Hergalant S, Rubio MT, D'Aveni M. Highly immunosuppressive myeloid cells correlate with early relapse after allogeneic stem cell transplantation. Exp Hematol Oncol. 2024 May 11;13(1):50. doi: 10.1186/s40164-024-00516-4. PMID 38734654